CLINICAL TRIAL: NCT01592877
Title: Clinical Test of Ultra-Wideband Non-contact Heart Rate and Breath Rate Monitor
Brief Title: A Comparative Study of the Performance of a New Type Non-contact Patient Monitor
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Holux Technology, Inc. (Industry)
Collaborators: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Holux_SKH01
Record Dates: First submitted 2012-05-04; First posted 2012-05-07 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Indication for Modification of Patient's Cardiopulmonary Status
Keywords: UWB; non-contact; patient monitor

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To verify the accuracy and reliability of the ultra wideband (UWB) non-contact breath rate and heart rate monitor, ICU bedside monitor is used as the gold standard.

DETAILED DESCRIPTION:
In this study, 50 volunteer patients are tested on the UWB non-contact breath rate and heart rate monitor. The testing time length for each patient is set to two hours. Subject is not to be restrained and nurse is allowed to take care the subject while testing. The breath rate and heart rate data will be analyzed for their accuracy against the MP60 (Philips) bedside monitor.

ELIGIBILITY:
Inclusion Criteria:

* conscious adult,
* > 18 years old

Exclusion Criteria:

* non-conscious,
* pregnant women,
* epilepsy patients,
* patients with heart pacemaker or ACIDS,
* patients on respirator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult, >18 years old.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2011-12; Primary Completion 2012-10 (Estimated); Study Completion 2012-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Che-Ming Chang, MD, Principal Investigator — Shin Kong Wu Ho-Su Memorial Hospital
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan